CLINICAL TRIAL: NCT05527119
Title: Phenotyping and Genotyping of Duffy Antigen
Acronym: DARC
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8543
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Plasmodium Vivax
Keywords: Malaria; Malaria, Vivax; PvDBP-DARC interaction; Plasmodium vivax; Duffy-negative; Duffy Binding Protein; PvDBP; Duffy Antigen Receptor for Chemokines
MeSH Terms: conditions — Malaria, Vivax; Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malaria remains the world's leading parasitic endemic. Almost half of the world's population lives in endemic areas. Many at-risk people in African countries remain without access to malaria control. Malaria kills approximately 400,000 people each year, most of whom are children under the age of 5 in Africa. Since 2005, an increasing number of Plasmodium vivax infections have been observed in Duffy-negative populations in South America and Africa, calling into question the essential role of the PvDBP-DARC interaction. The objective of the investigators is therefore to study and understand the invasion pathways used by Plasmodium vivax in Duffy-negative subjects.

ELIGIBILITY:
Inclusion Criteria:

* Major subjects
* with malaria and willing to have their blood samples analyzed for this research

Exclusion Criteria:

* Subjects refusing to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Major subjects with malaria and willing to have their blood samples analyzed for this research
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Number of blood samples tested (phenotype and genotype). | 2 months later

CONTACTS AND LOCATIONS:
Overall Officials: Didier MENARD, MD, PhD, Principal Investigator — Service Laboratoire de Parasitologie et Mycologie Médicale-PTM - CHU de Strasbourg - France
Locations (1):
- Service de Laboratoire de Parasitologie et Mycologie Médicale-PTM - CHU de Strasbourg - France, Strasbourg, France